CLINICAL TRIAL: NCT01973712
Title: Treatment of Periprosthetic Distal Femur Fractures: A Randomized Controlled Trial of Locking Plate Osteosynthesis Versus Retrograde Nailing
Brief Title: Periprosthetic Distal Femur Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPDF
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Periprosthetic Fractures; Distal Femur Fractures
MeSH Terms: conditions — Periprosthetic Fractures; Femoral Fractures, Distal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Locked Compression Plating (Experimental): A direct lateral approach to the distal femur will be employed utilizing minimally invasive and indirect reduction techniques. After fracture reduction is achieved with the use of intra-operative fluoroscopy, a locking plate will be provisionally implanted. Following confirmation of placement, definitive fixation will follow with multiple locking screws in the distal fragment and bicortical screw fixation proximally. A standard layered closure will follow
  Interventions: Procedure: Locked Compression Plating
- Retrograde Intramedullary Nailing (RIMN) (Experimental): The previous midline knee incision will be employed to access to the knee joint, allowing exposure of the femoral start point via the open box in the femoral component. Following reaming of the canal, an appropriately sized retrograde nail will be inserted. Intra-operative fluoroscopy will be used to confirm reduction. Both proximal and distal locking screws will be used to transfix the nail. A standard layered closure will follow.
  Interventions: Procedure: Retrograde Intramedullary Nailing (RIMN)

INTERVENTIONS:
Procedure: Locked Compression Plating
  Arms: Locked Compression Plating
Procedure: Retrograde Intramedullary Nailing (RIMN)
  Arms: Retrograde Intramedullary Nailing (RIMN)

SUMMARY:
A periprosthetic distal femur fracture is a fracture close to a knee implant. This type of fracture is often difficult to fix because of the close proximity of the two surgical implants which can sometimes interfere with proper bone healing. Improper healing can cause significant impairment and sometimes requires additional surgeries to correct the problem. Despite considerable interest and research put into developing techniques to repair this fracture surgeons do not know which is the best way to treat this type of fracture.

Our multicentre orthopaedic study group is conducting this study to compare two standard, but different treatments for periprosthetic distal femur fractures. One treatment consists of open surgery and the placement of a plate and screws along the side of the femur. The other consists of implanting an intramedullary nail in the femur.

The goal of this study is to directly compare the two treatments to see if one treatment results in better patient outcomes than the other.

ELIGIBILITY:
INCLUSION CRITERIA:

Age 18 years and older Displaced periprosthetic fracture of the distal femur Fracture amenable to both treatment groups, in the opinion of the investigator Knee prosthesis is well-fixed and non-stemmed Open box femoral component Provision of written informed consent

EXCLUSION CRITERIA:

Presence of an active infection around the fracture (soft tissue or bone) Open fracture Injury Severity Score (ISS) > 15 or any associated major injuries of the lower extremities Medical contraindication to surgery Pregnant women Likely problems, in the judgment of the investigators, with maintaining follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2014-05; Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) test | 3 months
  The TUG is a very simple timed test that was introduced in 1991 to measure mobility in the elderly. It involves documenting the time, in seconds, taken for subjects to rise from a standard arm chair, walk to a line on the floor 3 meters away, turn, return, and sit down again

SECONDARY OUTCOMES:
Rates of re-operation | 12 months

OTHER OUTCOMES:
Rates of malunion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Nauth, MD, FRCSC, Principal Investigator — Unity Health Toronto; Emil Schemitsch, MD, FRCSC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Department of Orthopaedic Surgery, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Claireaux HA, Searle HKC, Parsons NR, Griffin XL. Interventions for treating fractures of the distal femur in adults. Cochrane Database Syst Rev. 2022 Oct 5;10(10):CD010606. doi: 10.1002/14651858.CD010606.pub3. PMID 36197809